CLINICAL TRIAL: NCT05442684
Title: A Multicenter, Randomized, and Observer-blind Clinical Trial to Evaluate the Safety and Immunogenicity of Ad5-based COVID-19 Vaccine Against Coronavirus Variants in Adults (≥ 18 Years) Who Have Been Immunized With 2 Doses of mRNA Vaccines Plus One Dose of Booster AZD1222 Vaccine
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Ad5-vector Based Vaccine Against Coronavirus Variants in Adults (≥18 Years) Immunized With 2 Doses of mRNA Vaccines Plus One Dose of Booster AZD1222 Vaccine
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial protocol was not approved by the regulatory authorities.
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CTP-AD5NCOV/O-001
Record Dates: First submitted 2022-06-16; First posted 2022-07-05 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Subjects who have completed the primary mRNA vaccine immunizations and the 1st booster AZD1222 immunization for more than 6 months will be randomized to receive a 2nd booster dose of Ad5-nCoV/O, Ad5-nCoV/O-IH or mRNA-based COVID-19 vaccine in a ratio of 2:2:1.
Who Masked: Investigator
Masking Description: observer-blind clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ad5-nCoV/O group (Experimental)
  Interventions: Biological: Bivalent Recombinant COVID-19 Vaccine (Adenovirus Type 5 Vector)
- Ad5-nCoV/O-IH group (Experimental)
  Interventions: Biological: Bivalent Recombinant COVID-19 Vaccine (Adenovirus Type 5 Vector) for Inhalation
- mRNA-based COVID-19 vaccine group (Active Comparator)
  Interventions: Biological: mRNA-based COVID-19 vaccine

INTERVENTIONS:
Biological: Bivalent Recombinant COVID-19 Vaccine (Adenovirus Type 5 Vector) — Subjects who have completed the primary mRNA vaccine immunizations and the 1st booster AZD1222 immunization for more than 6 months will be randomized to receive a 2nd booster dose of Ad5-nCoV/O
  Arms: Ad5-nCoV/O group
Biological: Bivalent Recombinant COVID-19 Vaccine (Adenovirus Type 5 Vector) for Inhalation — Subjects who have completed the primary mRNA vaccine immunizations and the 1st booster AZD1222 immunization for more than 6 months will be randomized to receive a 2nd booster dose of Ad5-nCoV/O-IH
  Arms: Ad5-nCoV/O-IH group
Biological: mRNA-based COVID-19 vaccine — Subjects who have completed the primary mRNA vaccine immunizations and the 1st booster AZD1222 immunization for more than 6 months will be randomized to receive a 2nd booster dose of mRNA-based COVID-19 vaccine
  Arms: mRNA-based COVID-19 vaccine group

SUMMARY:
Subjects who have completed the primary mRNA vaccine immunizations and the 1st booster AZD1222 immunization for more than 6 months will be randomized to receive a 2nd booster dose of Ad5-nCoV/O, Ad5-nCoV/O-IH or mRNA-based COVID-19 vaccine in a ratio of 2:2:1.

DETAILED DESCRIPTION:
This is a multicenter, randomized, observer-blind, and parallel-controlled clinical study to evaluate the immune responses and safety profiles in adults (≥ 18 years) receiving investigational products (intramuscular injection or nebulized inhalation) ≥ 180 days after the immunization of 2 doses of BNT162b2 vaccines plus one dose of booster AZD1222 vaccine. This study will enroll about 30% participants aged 60 years and above.

Subjects who have completed the primary mRNA vaccine immunizations and the 1st booster AZD1222 immunization for more than 6 months will be randomized to receive a 2nd booster dose of Ad5-nCoV/O, Ad5-nCoV/O-IH or mRNA-based COVID-19 vaccine in a ratio of 2:2:1.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 years and above at the time of screening.
2. Received the 1st booster vaccination at least 180 days earlier.
3. Agree to attend all visits and sign the written informed consent form.

Exclusion Criteria:

1. Have a history of seizures, epilepsy, encephalopathy, psychosis.
2. History of severe anaphylaxis or allergy to any vaccine component.
3. Positive urine pregnancy test result, pregnant, lactating women.
4. Medical history of Guillain-Barré syndrome.
5. Have had asthma attacks within 2 years.
6. Have severe nasal or oral diseases, such as rhinitis (sinusitis), allergic rhinitis, oral ulcer, throat swelling, etc.
7. Bleeding disorder (e.g. protein S or factor deficiency, coagulopathy or platelet disorder).
8. Have chronic systematic infection or chronic obstructive pulmonary disease (COPD), etc.
9. Administration of immunoglobulins and/or any blood products within three months prior to the planned administration of the vaccine candidate.
10. Current diagnosis or receiving treatment for tuberculosis or cancer.
11. History of SARS-CoV-2 infection for less than 3 months.
12. Received or plan to receive any vaccines (licensed or investigational), within 14 days before and after study vaccination.
13. Have an axillary temperature of > 37.0℃.
14. Any other significant diseases, disorders or findings which may significantly increase the risk to the volunteer because of participation in the study, and affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of Ad5-nCoV/O or Ad5-nCoV/O-IH versus BNT162b2 as the 2nd booster dose. | Day 28 post vaccination
  The geometric mean titers (GMT) of anti-Omicron pseudovirus neutralizing antibody on Day 28 post vaccination in all participants

SECONDARY OUTCOMES:
Incidence of Adverse Reactions (ARs) | within 30 min post vaccination
  The incidence of adverse reactions (ARs) within 30 min post vaccination.
Incidence of Adverse Reactions (ARs) | within 14 days post vaccination
  The incidence of adverse reactions (ARs) within 14 days post vaccination
The incidence of AR and AE | within 28 days post vaccination
  The incidence of ARs/adverse events (AEs) within 28 days post vaccination.
Incidence of SAE | within 12 months post vaccination
  The incidence of serious adverse events (SAEs) and adverse events of special interest (AESIs) within 12 months post vaccination.
Immunogenicity of pseudovirus neutralizing antibody | on Day 14 and Day 28 post-vaccination
  The GMT, geometric mean increase fold (GMI) and sero-conversion rate (SCR) of anti-Omicron pseudovirus neutralizing antibody on Day 14 and Day 28 post-vaccination in all participants.
Immunogenicity of S-RBD IgG antibody | on Day 14 and Day 28 post-vaccination
  The geometric mean concentration (GMC), GMI and SCR of anti-Omicron S-RBD IgG antibody on Day 14 and Day 28 post-vaccination in all participants.
Immunogenicity of S-RBD serum IgA antibody | on Day 14 and Day 28 post-vaccination
  The GMT, GMI, and SCR of anti-Omicron S-RBD serum IgA antibody on Day 14 and Day 28 post-vaccination in all participants.
Immunogenicity of pseudovirus neutralizing antibody | on Month 3, Month 6, and Month 12 post-vaccination
  The GMT, GMI and SCR of anti-Omicron pseudovirus neutralizing antibody on Month 3, Month 6, and Month 12 post-vaccination in participants of the immunogenicity subgroup.
Immunogenicity of S-RBD IgG antibody | on Month 3, Month 6, and Month 12 post-vaccination
  The GMC, GMI and SCR of anti-Omicron S-RBD IgG antibody on Month 3, Month 6, and Month 12 post-vaccination in participants of the immunogenicity subgroup.
Immunogenicity of S-RBD serum IgA antibody | on Month 3, Month 6, and Month 12 post-vaccination
  The GMC, GMI and SCR of anti-Omicron S-RBD serum IgA antibody on Month 3, Month 6, and Month 12 post-vaccination in participants of the immunogenicity subgroup
Virological confirmed COVID-19 cases | from Day 14 post-vaccination
  The number of virological confirmed COVID-19 cases occurring from Day 14 post-vaccination in different vaccine groups.
Virological confirmed severe COVID-19 cases. | from Day 14 post-vaccination
  The number of virological confirmed severe COVID-19 cases occurring from Day 14 post-vaccination in different vaccine groups.
Virological confirmed asymptomatic COVID-19 cases | from Day 14 post-vaccination
  The number of virological confirmed asymptomatic COVID-19 cases occurring from Day 14 post-vaccination in different vaccine groups.
Immunogenicity of anti-Nucleocapsid antibody | before vaccination
  The GMT of anti-Nucleocapsid antibody before vaccination
Immunogenicity of saliva secretory IgA (SIgA) | on Day 14 and Day 28 post-vaccination
  The GMC, GMI, and SCR of saliva secretory IgA (SIgA) on Day 14 and Day 28 post-vaccination in participants of the immunogenicity subgroup.
The level and positive rate of interferon γ (IFN-γ) | on Day 14 and Day 28 after the 2nd booster dose
  The level and positive rate of interferon γ (IFN-γ) on Day 14 and Day 28 after the 2nd booster dose.
The neutralizing antibody against other VOCs or emerging variant(s). | on Day 28
  The neutralizing antibody on Day 28 against VOCs or other emerging variants.

IPD SHARING:
Plan to Share IPD: No